CLINICAL TRIAL: NCT05632796
Title: Can the Length of the Pfannenstiel Skin Incision be Adjusted According to the Fetal Head During Elective/Planned Cesarean Delivery?
Brief Title: Tailored Pfannenstiel Incision for Caesarean Delivery According to the Fetal Head Occipitofrontal Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Baris KAYA, Associate Professor, Near East University, Turkey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cesarean incision-1398
Record Dates: First submitted 2022-11-14; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Incision, Surgical; Cesarean Delivery Affecting Fetus; Pfannenstiel Incision Length; Fetal Occipitofrontal Diameter
Keywords: cesarean delivery; Pfannenstiel incision length; occipitofrontal diameter
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tailored pfannenstiel incision according to the fetal head OFD (Experimental): Pfannenstiel incision performed according to the occipitofrontal diameter of the fetal head
  Interventions: Procedure: Adjusting the Pfannenstiel skin incision according to the occipitofrontal diameter (OFD) of the fetal head.

INTERVENTIONS:
Procedure: Adjusting the Pfannenstiel skin incision according to the occipitofrontal diameter (OFD) of the fetal head. — All women will be subjected to regional spinal anesthesia. Pfannenstiel incision will be made according to the fetal occiputofrontal diameter, marked on the skin (Pfannenstiel incison with Kaya modification) Following blunt entry to the abdominal cavity, the uterine lower segment Kerr incision will be performed. Folllowing delivery of the baby, umblical cord will be cut and an arterial umblical cord blood sample will be taken. Placenta will be removed. 1st and 5th min. Apgar scores will be noted. Uterine incison will be sutured double-layer with 1 polyglactin 910 suture . Peritoneum and fascia, will be closed with 2-0 and 1 polyglactin 910 suture respectively. Skin incision will be sutured with continuous 3-0 rapid polyglactin 910 suture and measured with flexible ruler in centimeters following completing the skin incision closure.

SUMMARY:
The purpose of the study is whether the Pfannenstiel skin incision can be adjusted according to the occipitofrontal diameter (OFD) of the fetal head.

DETAILED DESCRIPTION:
Eligable nulliparous women delivered at term by elective cesarean section in which Pfannenstiel skin incision was performed according to the occipitofrontal diameter (OFD) of the fetal head were included. Non-vertex presentaions, all emergency cesarean sections, severe preclampsia, women in active phase of the first stage of labor and second stage of labor, placenta pervia and low lying placenta, multiple pregnancies, uncontrolled gestational diabetes mellitus were excluded.

ELIGIBILITY:
Inclusion Criteria:

* The women older than 18 years
* term nulliparous pregnancies (>37w)
* primary elective/planned Cesarean delivery
* fetuses with vertex presentations
* underwent spinal anesthesia

Exclusion Criteria:

* all emergency cesarean sections ( fetal distress, third trimester bleeding including abruption of placenta and placenta previa bleeding, arrest of labor in the second phase)
* cesarean delivery for severe preeclampsia
* cesarean delivery for non-vertex fetal presentations (breech and shoulder presentation)
* cesarean delivery for deflexion fetal head presentations (face and brow)
* cesarean delivery during active phase of the first stage of labor
* cesarean delivery for placenta previa or low-lying placenta,
* cesarean delivery for multiple pregnancies
* all cesarean deliveries with uncontrolled gestational or non-gestational diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 115 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Final Pfannenstiel incision length | up to 48 months
  Pfannenstiel skin incision length measured as milimetre (mm) which was performed according to the fetal occipitofrontal diameter measured with ultrasonography before delivery
difference between the initial and the Pfannenstiel incision length | up to 48 months
  difference between the initial incision which was adjusted according to the fetal occipitofrontal diameter and the final Pfannenstiel incision in millimetre(mm)
rate of extension of the Pfannensitel skin incision in the study population | up to 48 months
  percentage of patients who need of extension of the Pfannensitel skin incision in which the novel technique was performed

SECONDARY OUTCOMES:
duration of cesarean delivery | up to 48 months
  duration of surgery starts with from the skin incision ends with closing the skin measured with minute
time interval between uterine incision and fetal delivery | up to 48 months
  time interval between starting the Kerr uterine incision and delivery of the fetus measured with seconds
cut of the abdominal rectus muscle during delivery of the fetus | up to 48 months
  number of participants who need cut of the abdominal rectus muscle during delivery of the fetus
health evaluation of the newborn with Apgar scoring system | up to 48 months
  evaluation of the of the health of the newborn with 1. min and 5. min Apgar scoring system (1-10)
evaluation of the fetal acidosis by measuring the umbilical blood ph levels | up to 48 months
  evaluation of fetal acidosis with umbilical ph values (7.15-7.49), < 7.1 is accepted as fetal acidosis

CONTACTS AND LOCATIONS:
Overall Officials: baris kaya, Assos.Prof, Principal Investigator — Near East University Faculty of Medicine, Lefkosa-10 TRNC, Mersin, Turkey
Locations (1):
- Near East University, Obstetrics and Gynecology, Mersin, TRNC, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
we may share our data upon request

REFERENCES:
- [Derived] Kaya B, Ozay OE, Ozay AC, Tuten A. Can the Pfannenstiel skin incision length be adjusted according to the fetal head during elective cesarean delivery? Front Surg. 2023 Sep 26;10:1227338. doi: 10.3389/fsurg.2023.1227338. eCollection 2023. PMID 37829600